CLINICAL TRIAL: NCT05665816
Title: Results of the Treatment of Medium and Long de Novo and Restenotic Lesions in the Superficial Femoral Artery and/or Popliteal Artery With Primary or Salvage Pulsar® -18 t3 Stent
Acronym: T3PROJECT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Other Study IDs: IMIB-STN-2022-02
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Peripheral Artery Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Subjects with PAD treated with the PULSAR® -18 T3 Stent will be assessed for eligibility for the registry and consecutively included in the registry. Once informed consent is obtained, the required data will be collected.
  Interventions: Device: Stent PULSAR® -18 T3,

INTERVENTIONS:
Device: Stent PULSAR® -18 T3, — Post-authorization, prospective and multicenter registry to evaluate the clinical results of the PULSAR® -18 T3 stent, in the treatment of de novo or restenotic lesions of the superficial femoral and/or popliteal artery, primarily as salvage, in a population of patients residing in Spain and in "real life" conditions.

SUMMARY:
The purpose of this post-authorization registry is to describe the clinical outcomes of de novo and restenotic lesions in the superficial femoral and/or popliteal artery treated with the PULSAR® -18 T3 stent, implanted both primary and salvage.

DETAILED DESCRIPTION:
Post-authorization, prospective and multicenter registry to evaluate the clinical results of the PULSAR® -18 T3 stent, in the treatment of de novo or restenotic lesions of the superficial femoral and/or popliteal artery, primarily as salvage, in a population of patients residing in Spain and in "real life" conditions.

In this registry, data will be collected from approximately 100 consecutive patients who have been treated with the PULSAR® -18 T3 Stent.

Subjects with PAD treated with the PULSAR® -18 T3 Stent will be assessed for eligibility for the registry and will be consecutively included in the registry. Once informed consent is obtained, the required data will be collected.

ELIGIBILITY:
Inclusion Criteria:

I1. Patients with documented PAD from the AFS and/or AP, classified as having intermittent claudication or critical limb ischemia (CLI), with a Rutherford score between 3 and 5.

I2. Age ≥ 55 years. I3. The target lesion consists of one or multiple de novo or restenotic lesions > 5 cm.

I4. Adequate run-off distal circulation to the foot (at least one patent, pre-existing, or successfully restored native distal vessel before beginning treatment of the target lesion).

I5. Adequate in-flow defined as, stenosis ≤ 30% of the diameter (either pre-existing or successfully reestablished before starting treatment of the target lesion).

I6. CI signed and dated.

Exclusion Criteria:

E1. Failure to successfully cross the target lesion with a guidewire (successful crossing means that the tip of the guidewire is distal to the target lesion, without dissection or perforation that limits blood flow).

E2. Life expectancy < 12 months.

E3. Any contraindication to the use of antiplatelet therapy and/or heparin

E4. Acute or subacute thrombosis in the target vessel.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the statistical analyzes will be carried out in the group of patients who have the necessary data to evaluate the main objective. Secondary objectives will be analyzed using available data only (missing data imputation techniques will not be used).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
No device- or procedure-related mortality | Up to 24 months.
  Number of deaths
No major amputation of the treated limb | Up to 24 months.
  Number of amputations
No revascularization of the target lesion | Up to 24 months.
  Number of lesions not revascularized
Revascularization rate of the clinically indicated target lesion | Up to 24 months.
  Number of new intervention of the target lesion, indicated by symptomatology or by a decrease in ABI (Ankle Brachial Index) ≥ 20% or ≥ 0.15 compared to the ABI after the index procedure or, a PSVR (Pick Systolic Velocity Ratio) > 2.4 measured by DUS (Doppler Ultrasound)

SECONDARY OUTCOMES:
Serious Adverse Event Rates | Up to 24 months.
  Number of serious adverse events
Rate of success of the procedure | Up to 24 months.
  Number of Residual stenosis ≤ 50% by visual estimation
Primary patency | Up to 24 months.
  Absence of CD-TLR (clinically indicated TLR) and target lesion restenosis during follow-up, greater than 50% as determined by PSVR > 2.4 according to DUS (Doppler Ultrasound)
Assisted primary patency. | Up to 24 months.
  Patency of the target lesion after reoperation due to any reason, the lesion being patent at that time.
Secondary patency. | Up to 24 months.
  Patency of the target lesion after treatment of a (re)occlusion of the target lesion.
Rate of Clinical improvement (based on the Rutherford and WIfI classification) or absence of critical ischemia | Up to 24 months.
  Number of patients with maintained decrease of minus 1 degree in CR and exit from critical ischemia compared to baseline.
Rate of patients with major amputation of target limb | Up to 24 months.
  Number of surgical removal of the target limb:
  * Supracondylar amputation: amputation of the limb with the resection point above the knee.
  * Infracondylar amputation: amputation of the limb with the resection point below the knee.
Hemodynamic improvement | Up to 24 months.
  Ankle Brachial Index
Mortality from any cause | Up to 24 months.
  Number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cuenca Manteca, MD, Principal Investigator — Hospital Universitario Santa Lucía Murcia

IPD SHARING:
Plan to Share IPD: Undecided